CLINICAL TRIAL: NCT02435966
Title: Effectiveness of Dry Needling on the Upper Trapezius and the Levator Scapulae in Patients With Chronic Neck Pain: Randomized Clinical Trial
Brief Title: Dry Needling in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Gracia Gallego Sendarrubias, Fisioterapeuta, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University European of Madrid
Record Dates: First submitted 2015-03-27; First posted 2015-05-06 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Manual therapy + Dry needling (Experimental): Manual therapy + Dry needling: 2 sessions, after a 7 days interval
  Interventions: Device: Dry needling; Other: Manual therapy
- Manual therapy + Sham Dry needling (Other): Manual therapy + Sham Dry needling: after a 7 days interval
  Interventions: Device: Sham Dry needling; Other: Manual therapy
- Untreated control (No Intervention): Natural history of the condition

INTERVENTIONS:
Device: Dry needling — Dry needling of the most active trigger point either in the upper trapezius or the levator scapulae with 40mm x 0,32mm ener-qi guided needles (EQ1132)
  Arms: Manual therapy + Dry needling
Device: Sham Dry needling — Sham Dry needling with a retractile needle (Park Sham Placebo Acupuncture Device) of the most active trigger point either in the upper trapezius or the levator scapulae
  Arms: Manual therapy + Sham Dry needling
Other: Manual therapy — Standard manual therapy in the upper trapezius or the levator scapulae
  Arms: Manual therapy + Dry needling; Manual therapy + Sham Dry needling

SUMMARY:
The investigators study the efficacy of a combination of dry needling plus manual therapy against sham dry needling plus manual therapy in the treatment of chronic neck pain. The investigators identify the most active trigger point in the upper trapezius and levator scapulae and administer two treatments, with an interval of 7 days, with a follow up 30 days after the first intervention. The primary outcome is the Visual Analogue Scale of Pain. Secondary outcomes ar pressure pain threshold, Neck Disability Index (NDI) questionnaire and range of motion.

DETAILED DESCRIPTION:
A prospective single-blind randomized controlled trial, designed to assess the efficacy of dry needling in the treatment of chronic neck pain. The treatment regimes simulate the standard physiotherapy administered in real clinical settings. Patients in the intervention group receive a combination of manual therapy and dry needling (40mmx0,32 guided needles). There are two control groups. In the first one, patients receive a combination of manual therapy and sham dry needling. In the second control group, patients receive no treatment in order to assess the natural history of the disease.

Patients receive two treatment sessions with an interval of 7 days and are followed up after 30 days. The primary outcome is subjective pain assessed with a Visual Analogue Scale (VAS). Secondary outcomes are pressure pain threshold (assessed with a manual algometer), neck range of motion (assessed with a goniometer) and the Neck Disability Index (a standardized questionnaire). Measurements are taken pre and post-test after the first and the second treatment sessions, plus once more at the follow-up, except for the Neck Disability Index (only at the beginning and after the second treatment). In the non-treated group, patients were measured at the same time intervals.

The sample size was calculated to detect a VAS difference of 2 points, the minimally clinically important difference established in the literature. Then it was doubled in order to avoid possible dropouts. The trial takes place in a private practice in Madrid (Physios, c/Valverde 26). Patients are randomized by a computer program.

Patients are explored for active trigger points in the upper trapezius and the levator scapulae. They should meet the criteria of identification established by Travell & Simons in their Trigger point manual. The investigators also seek for trigger points following Travell & Simons' pain maps for these two muscles, where they identify five trigger point areas. The investigators select the most active, taking pressure pain threshold measurements of all the active trigger point, normalizing the values according to normal thresholds for each of the five areas in the two muscles. The normal thresholds were assessed in a pilot study with healthy patients. The investigators administer either dry or sham dry needling to the most active (the one with the lowest pain threshold) throughout the trial.

Dry needling is applied following Hong's technique with 40mmx0,32 guided needles, by a physiotherapist with 4 years of experience in the technique.

ELIGIBILITY:
Inclusion criteria

* Neck pain for at least three months (or more)
* An active trigger point in either the upper trapezius or the levator scapulae

Exclusion criteria

* Treatment for neck pain within the previous six months
* Neck Whiplash
* Fibromyalgia
* Infection in the area under treatment
* Pharmacological treatment with anti-coagulants
* Fear to needles
* Degenerative conditions
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

REFERENCES:
- [Derived] Gallego-Sendarrubias GM, Rodriguez-Sanz D, Calvo-Lobo C, Martin JL. Efficacy of dry needling as an adjunct to manual therapy for patients with chronic mechanical neck pain: a randomised clinical trial. Acupunct Med. 2020 Aug;38(4):244-254. doi: 10.1136/acupmed-2018-011682. Epub 2020 Mar 23. PMID 32202124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between May 2013 and June 2014 at Physios, a private physiotherapy practice in central Madrid (Spain)
Pre-assignment Details: No significant event here
Period: Overall Study
Arm/Group | Manual Therapy + Dry Needling | Manual Therapy + Sham Dry Needling | Untreated Control
Started | 47 | 54 | 30
First Intervention | 47 | 54 | 30
Second Intervention | 47 | 53 | 30
Follow-up | 47 | 53 | 30
Completed | 47 | 53 | 30
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Therapy + Dry Needling | Manual Therapy + Sham Dry Needling | Untreated Control | Total
Number analyzed (Participants) | 47 | 54 | 30 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.13 (7.64) | 34.64 (8.88) | 31.37 (9.33) | 34.62 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 16 | 80
  Male | 13 | 24 | 14 | 51
Visual Analogue Scale [Mean (Standard Deviation); unit: units on a scale] | 6.66 (1.37) | 6.17 (1.60) | 6.57 (1.33) | 6.44 (1.46)
Pressure Pain Threshold at the most active trigger point [Mean (Standard Deviation); unit: kg/cm2] | 1.75 (0.37) | 1.88 (0.52) | 1.83 (0.43) | 1.82 (0.45)
Range of Motion (Neck): Rotation Left [Mean (Standard Deviation); unit: degrees] | 71.78 (17.73) | 73.81 (11.82) | 78.20 (11.21) | 74.09 (14.23)
Range of Motion (Neck): Rotation Rigth [Mean (Standard Deviation); unit: degrees] | 74.27 (18.10) | 74.60 (15.31) | 78.20 (11.21) | 76.24 (15.49)
Range of Motion (Neck): Flexion [Mean (Standard Deviation); unit: degrees] | 67.89 (13.53) | 69.24 (11.05) | 65.96 (8.82) | 68.00 (11.56)
Range of Motion (Neck): Extension [Mean (Standard Deviation); unit: degrees] | 52.31 (14.56) | 55.67 (11.54) | 59.66 (9.30) | 55.38 (12.50)
Range of Motion (Neck): Inclination Left [Mean (Standard Deviation); unit: degrees] | 53.63 (10.83) | 55.43 (10.99) | 52.43 (8.44) | 54.09 (10.39)
Range of Motion (Neck): Inclination Rigth [Mean (Standard Deviation); unit: degrees] | 47.72 (14.28) | 49.03 (13.09) | 45.63 (6.78) | 47.77 (12.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores on the Visual Analog Scale (VAS: 0-10) After 30 Days
Description: The Visual Analogue Scale is a validated, self-reported instrument to assess pain, with scores ranging from 0 (no pain) to 10 (maximum pain). We assess the change in chronic neck pain after 30 days, after to interventions in days 1 and 7) as compared to the baseline VAS
Time Frame: Pre-intervention (Day 1); After 1st intervention (Day 1); after 2nd intervention (7 days later); after followup (30 days later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual Therapy + Dry Needling | Manual Therapy + Sham Dry Needling | Untreated Control
Number analyzed (Participants) | 47 | 54 | 30
units on a scale | 1.77 (1.38) | 3.34 (1.92) | 8.83 (1.64)

2. Secondary Outcome: Change in the Pressure Pain Threshold Measured by Algometer
Description: Measured by algometer, with the standard measurement procedure
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Secondary Outcome: Change in the Cervical Range of Motion Measured by Goniometer
Description: Measured by goniometer, with the standard measurement procedure
Time Frame: as for outcome 1
Reporting Status: Not Posted

4. Secondary Outcome: Change in the Neck Disability Index Questionnaire
Time Frame: Pre-intervention (Day 1); after 2nd intervention (7 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days, from intervention 1 to follow-up
Arm/Group | Manual Therapy + Dry Needling | Manual Therapy + Sham Dry Needling | Untreated Control
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/54 | 0/30
Other Adverse Events (participants affected / at risk) | 0/47 | 0/54 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No